CLINICAL TRIAL: NCT01753323
Title: A Proof-of-concept, Open Label Study to Assess Efficacy, Safety, Tolerability and Pharmacokinetics of KAF156 in Adult Patients With Acute, Uncomplicated Plasmodium Falciparum or Vivax Malaria Mono-infection
Brief Title: Efficacy, Safety, Tolerability and Pharmacokinetics of KAF156 in Adult Patients With Acute, Uncomplicated Plasmodium Falciparum or Vivax Malaria Mono-infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CKAF156X2201
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Malaria
Keywords: acute malaria, KAF156
MeSH Terms: conditions — Malaria; Acute malaria | interventions — ganaplacide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 - Cohort 1: P. vivax: KAF156 400mg QD (Experimental): Participants with Plasmodium vivax malaria received KAF156 400 mg once a day for three days.
  Interventions: Drug: KAF156
- Part 1 - Cohort 2: P. falciparum: KAF156 400mg QD (Experimental): Participants with Plasmodium falciparum malaria received KAF156 400mg once a day for three days.
  Interventions: Drug: KAF156
- Part 2 - Cohort 3: P. falciparum: KAF156 800mg single dose (Experimental): Participants with Plasmodium falciparum malaria received a single dose of KAF156 800mg.
  Interventions: Drug: KAF156

INTERVENTIONS:
Drug: KAF156 — KAF156 was supplied as tablets for oral use.

SUMMARY:
This study will assess efficacy, safety , tolerability and PK in uncomplicated adult malaria patients with P. vivax or P. falciparum infection after 3 day dosing with KAF156 at 400 mg/day (Part 1) and single dosing with KAF156 at 800mg (Part 2)

ELIGIBILITY:
Inclusion Criteria:

-Male and female patients aged 20 to 60 years;Presence of mono-infection of P. falciparum or P. vivax; Weight between 40 kg to 90 kg.

Exclusion Criteria:

* Patients with signs and symptoms of severe/complicated malaria
* Infection with more than one parasite species
* Women of child-bearing potential; pregnant or nursing women
* Those who have taken any anti-malarial treatment in the preceding 14 days or other investigational drugs within 30 days or 5 half-lives

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Thailand (3):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Si Sa Ket
  - Novartis Investigative Site, Tak
- Novartis Investigative Site, Hanoi, Vietnam

REFERENCES:
- [Derived] White NJ, Duong TT, Uthaisin C, Nosten F, Phyo AP, Hanboonkunupakarn B, Pukrittayakamee S, Jittamala P, Chuthasmit K, Cheung MS, Feng Y, Li R, Magnusson B, Sultan M, Wieser D, Xun X, Zhao R, Diagana TT, Pertel P, Leong FJ. Antimalarial Activity of KAF156 in Falciparum and Vivax Malaria. N Engl J Med. 2016 Sep 22;375(12):1152-60. doi: 10.1056/NEJMoa1602250. PMID 27653565

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment of P. vivax malaria patients (Cohort 1) began first. Then the falciparum cohort began enrollment after four vivax patients had completed their dosing. Cohort 3 was enrolled after the completion of an interim analysis of safety, tolerability and efficacy data of seven completed patients in the second cohort of Part 1.
Period: Overall Study
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Started | 11 | 10 | 22
Pharmacodynamic (PD) Set | 10 | 10 | 21
Pharmacokinetic(PK) Set | 10 | 10 | 21
Safety Set | 11 | 10 | 22
Intent-to-treat Analysis Set | 11 | 10 | 22
Completed | 10 | 10 | 13
Not Completed | 1 | 0 | 9
Not completed — Lack of Efficacy | 0 | 0 | 8
Not completed — Protocol deviation | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose | Total
Number analyzed (Participants) | 11 | 10 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.1 (8.42) | 36.7 (10.90) | 28.9 (7.00) | 31.2 (8.77)
Sex/Gender, Customized [Number; unit: Participants] — Males only
  Participants | 11 | 10 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Time to Parasite Clearance
Description: Parasite clearance was determined by assessing the parasite count in blood, using thin film, thick film and blood density assessments.
Time Frame: Day 5
Population: Pharmacodynamic (PD) analysis set for Cohorts 1, 2 and 3: The PD set included all participants who received at least one dose of study medication except for 1 participant from Cohort 1, who was excluded due to a protocol deviation, and 1 participant from Cohort 3, who was withdrawn on Day 1.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Number analyzed (Participants) | 10 | 10 | 21
Hours | 23.63 [16.00 to 30.02] | 44.97 [36.25 to 47.98] | 48.75 [42.00 to 53.95]

2. Primary Outcome: 28-day Cure Rate - Part 2
Description: 28-day cure rate was defined as the percentage of participants with blood parasite count of zero after 28 days of treatment.
Time Frame: Day 28
Population: Intent-to-treat analysis set: the intent-to-treat analysis set included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Number analyzed (Participants) | 22
Percentage of participants | 63.6

3. Secondary Outcome: Area Under the Curve (AUC)0-24h - Part 1
Description: AUC0-24h was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose. The 24h sampling of first post dose was taken before the second dose. On Day 3, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Days 1 and 3
Population: Pharmacokinetic (PK) analysis set for Cohorts 1 and 2: The PK set included all participants who received at least one dose of study medication except for 1 participant from Cohort 1, who was excluded due to a protocol deviation.
Measure: Mean (Standard Deviation); unit: (hr*ng/mL)
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD
Number analyzed (Participants) | 10 | 10
(hr*ng/mL)
  Day 1 | 9470 (2140) | 10100 (2440)
  Day 3 | 20200 (3730) | 21700 (6630)

4. Secondary Outcome: Maximum Concentration (Cmax) - Part 1
Description: Cmax was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose. The 24h sampling of first post dose should be taken before the second dose. On Day 3, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Days 1 and 3
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD
Number analyzed (Participants) | 10 | 10
ng/mL
  Day 1 | 795 (182) | 856 (158)
  Day 3 | 1440 (299) | 1620 (384)

5. Secondary Outcome: Time to Maximum Concentration (Tmax) - Part 1
Description: Tmax was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose. The 24h sampling of first post dose should be taken before the second dose. On Day 3, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Days 1 and 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD
Number analyzed (Participants) | 10 | 10
hour
  Day 1 | 3.00 [2.00 to 6.00] | 3.00 [1.00 to 4.03]
  Day 3 | 3.00 [2.00 to 5.98] | 2.52 [2.00 to 3.02]

6. Secondary Outcome: Area Under the Curve (AUC)Last - Part 1
Description: AUClast was analyzed using parent drug in plasma samples. On Day 3, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Day 3
Population: as for outcome 3
Measure: Mean (Standard Error); unit: hr*ng/mL
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD
Number analyzed (Participants) | 10 | 10
hr*ng/mL | 55800 (12800) | 54300 (22500)

7. Secondary Outcome: Area Under the Curve (AUC)Inf - Part 1
Description: AUCinf was analyzed using parent drug in plasma samples. On Day 3, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD
Number analyzed (Participants) | 10 | 10
hr*ng/mL | 58300 (14500) | 56700 (24800)

8. Secondary Outcome: Half-life (T1/2) - Part 1
Description: T1/2 was analyzed using parent drug in plasma samples. On day 3, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD
Number analyzed (Participants) | 10 | 10
hr | 39.0 (7.40) | 40.8 (8.37)

9. Secondary Outcome: Clearance (CL/F ) - Part 1
Description: CL/F was analyzed using parent drug in plasma samples. On day 3, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD
Number analyzed (Participants) | 10 | 10
L/hr | 20.4 (4.04) | 19.7 (5.12)

10. Secondary Outcome: Apparent Volume of Distribution During the Terminal Elimination Phase Following Extravascular Administration (Vz/F) - Part 1
Description: Vz/F was analyzed using parent drug in plasma samples. On Day 3, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD
Number analyzed (Participants) | 10 | 10
Liters | 1150 (286) | 1140 (288)

11. Secondary Outcome: Accumulation Ratio (Racc) (=AUC0-24h, day3/AUC0-24h, day1) - Part 1
Description: Racc was analyzed using parent drug in plasma samples. On day 3, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD
Number analyzed (Participants) | 10 | 10
ratio | 2.16 (0.256) | 2.15 (0.384)

12. Secondary Outcome: AUC0-24h - Part 2
Description: AUC0-24h was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose.
Time Frame: Day 1
Population: Pharmacokinetic (PK) analysis set analysis set for Cohort 3: The PK set for Cohort 3 included participants who received at least one dose of study medication except for 1 participant who was withdrawn on Day 1 and 3 participants who vomited before 3 hours.
Measure: Mean (Standard Error); unit: hr*ng/mL
Arm/Group | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Number analyzed (Participants) | 18
hr*ng/mL | 21700 (5680)

13. Secondary Outcome: AUC0-48h - Part 2
Description: AUC0-48h was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Day 1
Population: as for outcome 12
Measure: Mean (Standard Error); unit: hr*ng/mL
Arm/Group | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Number analyzed (Participants) | 18
hr*ng/mL | 33600 (9150)

14. Secondary Outcome: AUClast - Part 2
Description: AUClast was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose
Time Frame: Day 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Number analyzed (Participants) | 18
hr*ng/mL | 54900 (16600)

15. Secondary Outcome: AUCinf - Part 2
Description: AUCinf was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose
Time Frame: Day 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Number analyzed (Participants) | 18
hr*ng/mL | 58300 (18600)

16. Secondary Outcome: Cmax - Part 2
Description: Cmax was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose.
Time Frame: Day 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Number analyzed (Participants) | 18
ng/mL | 1800 (404)

17. Secondary Outcome: Tmax - Part 2
Description: Tmax was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose.
Time Frame: Day 1
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Number analyzed (Participants) | 18
hours | 3.52 [2.00 to 11.6]

18. Secondary Outcome: T1/2 - Part 2
Description: T1/2 was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Day 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Number analyzed (Participants) | 18
hours | 48.7 (7.85)

19. Secondary Outcome: CL/F - Part 2
Description: CL/F was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Day 1
Population: Pharmacokinetic (PK) analysis set analysis set for Cohort 3: The PK set for Cohort 3 included participants who received at least one dose of study medication except for 1 participant who was withdrawn on Day 1 and 3 participants who who vomited before 3 hours.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Number analyzed (Participants) | 18
L/hr | 15.1 (4.85)

20. Secondary Outcome: Vz/F - Part 2
Description: Vz/F was analyzed using parent drug in plasma samples. On Day 1, samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, and 192 hours post dose.
Time Frame: Day 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Number analyzed (Participants) | 18
Liters | 1030 (264)

ADVERSE EVENTS:
Arm/Group | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/22
Other Adverse Events (participants affected / at risk) | 5/11 | 8/10 | 22/22
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Cohort 1: P. Vivax: KAF156 400mg QD (N=11) | Part 1 - Cohort 2: P. Falciparum: KAF156 400mg QD (N=10) | Part 2 - Cohort 3: P. Falciparum: KAF156 800mg Single Dose (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 7
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 13
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 3 | 14
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 1 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1 | 6
Fatigue (General disorders) | 0 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 4
Malaria (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 3
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 3
Eosinophil count increased (Investigations) | 1 | 0 | 0
Monocyte count decreased (Investigations) | 0 | 1 | 0
Monocyte count increased (Investigations) | 2 | 0 | 0
Thyroxine free increased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 2
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.